CLINICAL TRIAL: NCT05092113
Title: The Efficacy and Safety of a Compound Glutamine Capsule in the Primmary Prevention of Chemotherapy-induced Mucositis in Patients With Gastrointestinal Tumors: a Prospective, Randomized, Controlled, Double-blind, Phase III Clinical Study
Brief Title: The Efficacy and Safety of a Compound Glutamine Capsule in the Primary Prevention of Chemotherapy-induced Mucositis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meng Qiu (Other)
Responsible Party: Sponsor-Investigator, Meng Qiu, professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-615
Record Dates: First submitted 2021-09-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Mucositis; Chemotherapeutic Toxicity
Keywords: Chemotherapeutic Toxicity
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): a compound glutamine capsule was taken orally in the first cycle of chemotherapy, and a compound glutamine capsule simulated placebo was taken in the second cycle of chemotherapy. All patients take drugs orally on the first day of each cycle of chemotherapy, 3 tablets 3 times a day, and the course of the treatment was 3 weeks.
  Interventions: Drug: a compound glutamine capsule/a compound glutamine capsule simulated placebo
- Group B (Experimental): in the first cycle of chemotherapy, a compound glutamine capsule simulated placebo was given ,and in the second cycle, a compound glutamine capsule was taken at the same time of chemotherapy. All patients take orally from the first day of chemotherapy, 3 times a day after meals, 3 tablets each time, and the course of treatment was 3 weeks.
  Interventions: Drug: a compound glutamine capsule/a compound glutamine capsule simulated placebo

INTERVENTIONS:
Drug: a compound glutamine capsule/a compound glutamine capsule simulated placebo — A compound glutamine capsule/a compound glutamine capsule simulated placebo was taken orally from the first day of chemotherapy, orally 3 times a day after meals, 3 tablets each time, the course of treatment is 3 weeks.

SUMMARY:
Chemotherapy regimens not only improve the survival of patients with gastric cancer and colorectal cancer, but also cause obvious adverse reactions of digestive tract, such as chemotherapy-induced oral mucositis, abdominal pain, diarrhea, constipation and so on. These adverse reactions seriously affect the patients' quality of life and the efficacy of chemotherapy. Glutamine is a conditionally essential amino acid in the human body. Previous studies have shown that oral glutamine can help to keep the integrity of mucosal epithelium during chemotherapy and reduce the gastrointestinal side effects caused by chemotherapy. The addition of glutamine to parenteral nutrition can better maintain nitrogen balance and reduce the incidence of infection-related complications. A compound glutamine capsule, composed of L-glutamine and the traditional Chinese herbal formula Si-Jun-Zi-Tang which composed of ginseng, Atractylodes macrocephala, Poria cocos and licorice, has been widely used in China for 23 years to treat many types of gastrointestinal diseases, including gastrointestinal reactions induced by radiotherapy and chemotherapy, ulcerative colitis, irritable bowel syndrome. However, so far, only a small sample of clinical trials have explored the role of glutamine in chemical mucositis, and there is a lack of prospective randomized controlled clinical trials to further verify its value in the prevention and treatment of chemical mucositis. The purpose of this study is to observe the efficacy and safety between a compound glutamine capsule and placebo in the prevention of chemotherapy-induced mucositis in patients with gastric cancer and colorectal cancer in a prospective, randomized, double-blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Sex: Male or female
* Pathologically confirmed gastric adenocarcinoma or colorectal adenocarcinoma.
* Patients are ready to receive chemotherapy regimens containing platinum or irinotecan (targeted therapy could be used at the same time). Patients have not received any anti-cancer treatment before.
* patients are planned to receive the same chemotherapy regimen at least 2 cycles
* A baseline Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate haematopoietic function of bone marrow: neutrophils≥1.5x109 / L, platelets≥75x109 / L; normal liver and kidney function: TBIL≤ 1 upper limit of normal (ULN); ALT and AST ≤2.5 ULN; creatinine≤1.5 ULN.

Exclusion Criteria:

* (Patient-Generated Subjective Global Assessment, PG-SGA)>9 or severe malnutrition (weight loss > 10% or serum albumin < 30 g/L or body mass index < 18.5 kg/m2);
* Patients with severe heart, lung and brain diseases; chronic hepatitis infection, liver cirrhosis, chronic nephritis, kidney dysfunction, etc;
* Patients with infection-related fever;
* Patients who are known to be allergic or intolerant to any of the ingredients used in the study;
* Patients with long-term chronic diarrhea, abdominal pain, constipation or other digestive tract diseases; patients with gastrointestinal symptoms before chemotherapy (≥grade 2 NCI-CTCAE, version 4.0);
* Synchronously receive other treatments that may cause diarrhea, such as radiotherapy;
* Patients who take drugs for microecological regulation of digestive tract such as Combined Bifidobacterium, ChangTai oral liquid, etc;
* Patients take traditional Chinese medicine or antibiotics;
* Unable to understand and sign the informed consent form;
* participants in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of chemotherapy-induced diarrhea ≥ grade 1 | up to 3 weeks
  Overall incidence of chemotherapy-induced diarrhea ≥ grade 1 (according to National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0)

SECONDARY OUTCOMES:
Overall incidence of gastrointestinal adverse events except diarrhea ≥ grade 1 | up to 3 weeks
  Overall incidence of gastrointestinal adverse events except diarrhea ≥ grade 1 (including oral mucositis, nausea, vomiting, abdominal pain, stomachache, and other types, according to National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0)
Overall incidence of grade 3/4 gastrointestinal adverse events | up to 3 weeks
  Overall incidence of grade 3/4 gastrointestinal adverse events according to National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0

OTHER OUTCOMES:
Changes of scores of Quality of Life Questionare-Core 30 of the European Organization for Research and Treatment of Cancer of patients between interventional group and control group before and after this cycle of chemotherapy | an average of 3 weeks
  Changes of scores of Quality of Life Questionare-Core 30 of the European Organization for Research and Treatment of Cancer of patients between interventional group and control group before and after this cycle of chemotherapy
Changes of fecal flora and enteritis-associated inflammatory factors | an average of 3 weeks
  find the differences in the composition structure of the microbial community in the feces sample by 16SrDNA amplification techniques.Detect changes of calprotectin in patients in feces.

CONTACTS AND LOCATIONS:
Locations (1):
- Meng Qiu, Sichuan, China